CLINICAL TRIAL: NCT07194798
Title: A Prospective Randomized Trial Comparing the Posterior Pericardial Window Versus Retro-Cardiac Drain for the Prevention of Postoperative Atrial Fibrillation and Pericardial Complications Following CABG
Brief Title: Drainage Technique in CABG
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Saad Abdelhamid, Principal Investigator, Assiut University
Other Study IDs: Drainage technique in CABG
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: CABG; Atrial Fibrillation (AF)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: 61 patients undergoing CABG will have a posterior pericardial window created for drainage.: Based on determining the main outcome variable, the estimated minimum required sample size is 122 patients (61 patients in each group).
  * Group I (Posterior Pericardial Window group): 61 patients undergoing CABG will have a posterior pericardial window created for drainage.
  * Group II (Retro-cardiac Drain group): 61 patients undergoing CABG will receive a retro-cardiac drain for pericardial drainage.
- Group 2 : 61 patients undergoing CABG will receive a retro-cardiac drain for pericardial drainage.: Based on determining the main outcome variable, the estimated minimum required sample size is 122 patients (61 patients in each group).
  * Group I (Posterior Pericardial Window group): 61 patients undergoing CABG will have a posterior pericardial window created for drainage.
  * Group II (Retro-cardiac Drain group): 61 patients undergoing CABG will receive a retro-cardiac drain for pericardial drainage.

SUMMARY:
aims to compare the efficacy of the posterior pericardial window versus retro-cardiac drain in preventing postoperative atrial fibrillation and pericardial complications following CABG, while assessing their impact on hospital and ICU stay, pericardial effusions, re exploration for bleeding, post-operative blood transfusions, and mortality.

DETAILED DESCRIPTION:
Coronary artery bypass grafting (CABG) is a cornerstone in the management of advanced coronary artery disease, yet it carries a notable risk of postoperative complications. Among these, postoperative atrial fibrillation (POAF) is particularly common, affecting up to 40% of patients and contributing to increased morbidity, prolonged ICU and hospital stays, and elevated healthcare costs.

Pericardial effusion and tamponade are also frequent sequelae after CABG operation, often exacerbating the risk of POAF and necessitating re-intervention. Traditionally, retro-cardiac drains have been used to evacuate pericardial fluid, but their efficacy in preventing effusion-related complications is limited.

The posterior pericardial window (PPW) technique has emerged as a promising alternative, offering improved drainage and reduced incidence of POAF, early and late pericardial effusion, and tamponade. Studies have shown that PPW may also shorten ICU and hospital stays, reduce pleural effusion, and lower the need for revision surgery due to bleeding.

Despite encouraging data, randomized trials directly comparing PPW and retro-cardiac drains remain scarce. This study aims to fill that gap by evaluating the effectiveness of PPW versus retro-cardiac drain in preventing postoperative atrial fibrillation and pericardial complications following CABG, with secondary outcomes including pleural effusion, ICU/hospital stay duration, revision surgery, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18 and above) scheduled for elective, first-time coronary artery bypass grafting (CABG).
* Patients with preserved left ventricular function (ejection fraction ≥ 35%).
* Ability to provide informed consent and comply with follow-up protocols.
* No prior history of atrial fibrillation or other significant arrhythmias.

Exclusion Criteria:

* Patients undergoing combined cardiac procedures (e.g., valve repair or replacement).
* Emergency CABG cases or re-operations.
* Known bleeding disorders or ongoing anticoagulation therapy that cannot be paused.
* Severe pericardial adhesions or anatomical abnormalities preventing safe creation of a posterior pericardial window.
* Chronic pulmonary disease or pleural pathology that may interfere with drainage assessment.
* Patients with active infections or systemic inflammatory conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients scheduled to undergo elective, first-time, isolated coronary artery bypass grafting (CABG) surgery via median sternotomy. Eligible participants will be hemodynamically stable and able to provide informed consent prior to enrollment. Patients will be randomized intraoperatively to receive either a posterior pericardial window or a retro-cardiac drain for postoperative management.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative atrial fibrillation and pericardial complications | During hospitalization and up to 3 months after surgery
  Postoperative atrial fibrillation will be detected by continuous ECG monitoring during hospitalization. Pericardial complications, including early and late pericardial effusion, cardiac tamponade, and pleural effusion, will be assessed using echocardiography. The outcome will be reported as the number and percentage of participants experiencing any of these events.

SECONDARY OUTCOMES:
Postoperative clinical outcomes (ICU stay, hospital stay, revision surgery, and in-hospital mortality) | From surgery until hospital discharge (up to 30 days)
  Postoperative outcomes will include:
  Length of ICU stay and total hospital stay (measured in days from surgery until discharge).
  Requirement for revision surgery due to bleeding (documented from operative and postoperative records).
  All-cause in-hospital mortality (death from any cause during index hospitalization).
  These outcomes will be reported as duration in days and/or number and percentage of participants, as appropriate.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aranki SF, Shaw DP, Adams DH, Rizzo RJ, Couper GS, VanderVliet M, Collins JJ Jr, Cohn LH, Burstin HR. Predictors of atrial fibrillation after coronary artery surgery. Current trends and impact on hospital resources. Circulation. 1996 Aug 1;94(3):390-7. doi: 10.1161/01.cir.94.3.390. PMID 8759081
- [Background] Kalavrouziotis D, Buth KJ, Ali IS. The impact of new-onset atrial fibrillation on in-hospital mortality following cardiac surgery. Chest. 2007 Mar;131(3):833-839. doi: 10.1378/chest.06-0735. PMID 17356100
- [Background] Almassi GH, Schowalter T, Nicolosi AC, Aggarwal A, Moritz TE, Henderson WG, Tarazi R, Shroyer AL, Sethi GK, Grover FL, Hammermeister KE. Atrial fibrillation after cardiac surgery: a major morbid event? Ann Surg. 1997 Oct;226(4):501-11; discussion 511-3. doi: 10.1097/00000658-199710000-00011. PMID 9351718
- [Background] Mathew JP, Fontes ML, Tudor IC, Ramsay J, Duke P, Mazer CD, Barash PG, Hsu PH, Mangano DT; Investigators of the Ischemia Research and Education Foundation; Multicenter Study of Perioperative Ischemia Research Group. A multicenter risk index for atrial fibrillation after cardiac surgery. JAMA. 2004 Apr 14;291(14):1720-9. doi: 10.1001/jama.291.14.1720. PMID 15082699
- [Background] Maisel WH, Rawn JD, Stevenson WG. Atrial fibrillation after cardiac surgery. Ann Intern Med. 2001 Dec 18;135(12):1061-73. doi: 10.7326/0003-4819-135-12-200112180-00010. PMID 11747385
- [Background] Xiong T, Pu L, Ma YF, Zhu YL, Li H, Cui X, Li YX. Posterior pericardiotomy to prevent new-onset atrial fibrillation after coronary artery bypass grafting: a systematic review and meta-analysis of 10 randomized controlled trials. J Cardiothorac Surg. 2021 Aug 14;16(1):233. doi: 10.1186/s13019-021-01611-x. PMID 34391454
- [Background] Ranjan R, Kapetanakis S, Chandrasekaran V, Kaba RA, Momin AU. Posterior Pericardial Window and a Single Pleural Drain: A Dual Defence Against Post-CABG Pericardial Effusion and Atrial Fibrillation. Ther Clin Risk Manag. 2025 Apr 15;21:481-487. doi: 10.2147/TCRM.S521874. eCollection 2025. PMID 40255667